CLINICAL TRIAL: NCT06420388
Title: Efficacy of 2% Lidocaine Gel in Reducing Postoperative Pain and Analgesic Consumption Following Haemorrhoidectomy: A Randomized, Double-Blind, Controlled Trial
Brief Title: 2% Lidocaine Gel in Reducing Postoperative Pain Following Haemorrhoidectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: E-DA Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMRP28112N
Record Dates: First submitted 2024-05-12; First posted 2024-05-20 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Surgery; Pain, Postoperative
Keywords: hemorrhoids; pain management
MeSH Terms: conditions — Pain, Postoperative; Hemorrhoids; Agnosia

STUDY DESIGN:
Intervention Model Description: This study is a single-center, randomized, double-blind, controlled clinical trial comparing the efficacy of 2% lidocaine gel versus a non-anaesthetic lubricant gel control in reducing postoperative pain and analgesic consumption following haemorrhoidectomy. Patients were randomly assigned in a 1:1 ratio to either the intervention group receiving 5 mL 2% lidocaine gel three times per day postoperatively or the control group receiving 5 mL of a non-anaesthetic water-based lubricant gel.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study employed a double-blind masking approach to minimize potential bias. Patients, surgeons, and outcome assessors were blinded to treatment allocation. The randomization scheme was generated by a third party not involved in patient care, and sealed envelopes containing the allocation were opened only after the haemorrhoidectomy procedure was completed. The study gels were packaged identically to maintain blinding. Unblinding occurred only after data analysis was completed. This double-blind design ensured that knowledge of treatment allocation did not influence postoperative care, patient-reported pain scores, or the assessment of outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine Gel (Experimental): Description: Patients in this group received 5 mL of 2% lidocaine gel applied to the perianal region three times per day postoperatively. The gel was self-administered by the patient or applied by a nurse if the patient was unable to do so. Treatment continued for 7 days after the haemorrhoidectomy procedure.
  Arm Sample Size: 200
  Interventions: Drug: 2% Lidocaine Gel; Drug: Standard Postoperative Analgesics
- Controlled (Placebo Comparator): Description: Patients in this group received 5 mL of a non-anaesthetic, water-based lubricant gel (K-Y gel) applied to the perianal region three times per day postoperatively. The gel was self-administered by the patient or applied by a nurse if the patient was unable to do so. Treatment continued for 7 days after the haemorrhoidectomy procedure. This group served as a control to compare the efficacy of 2% lidocaine gel in reducing postoperative pain and analgesic consumption.
  Arm Sample Size: 200
  Interventions: Drug: Water-based Lubricant Gel (K-Y Gel); Drug: Standard Postoperative Analgesics

INTERVENTIONS:
Drug: 2% Lidocaine Gel — The intervention group received 5 mL of 2% lidocaine gel applied topically 3 times per day after undergoing Ferguson hemorrhoidectomy surgery.
  The control group received 5 mL of a non-anesthetic water-based lubricant gel applied topically 3 times per day after surgery.
  The application of the gels began immediately after surgery and continued for the postoperative period evaluated in the study.
  Both groups received standard postoperative analgesics (acetaminophen, celecoxib, Dynastat/parecoxib as needed) in addition to the topical gel applications.
  Arms: Lidocaine Gel
Drug: Water-based Lubricant Gel (K-Y Gel) — The intervention group received 5 mL of mL of a non-anesthetic water-based lubricant gel (K-Y gel) applied topically 3 times per day after undergoing Ferguson hemorrhoidectomy surgery.
  Arms: Controlled
Drug: Standard Postoperative Analgesics — Acetaminophen (Paracetamol)
  Dosage: 500 mg per tablet Frequency: Every 6 hours Route: Oral
  Acetaminophen is a common over-the-counter pain reliever and fever reducer. It works by blocking the production of prostaglandins, which are responsible for causing pain and inflammation.
  Celecoxib
  Dosage: 200 mg per tablet Frequency: Every 12 hours Route: Oral
  Celecoxib is a nonsteroidal anti-inflammatory drug (NSAID) that specifically inhibits the cyclooxygenase-2 enzyme. By reducing the production of prostaglandins, celecoxib helps alleviate pain and inflammation.
  Dynastat (Parecoxib)
  Dosage: 40 mg per injection Frequency: Every 12 hours as needed for poorly controlled pain Route: Intravenous

SUMMARY:
The study is a randomized, double-blind, controlled trial evaluating the efficacy of 2% lidocaine gel in reducing postoperative pain and analgesic consumption after haemorrhoidectomy. 222 patients undergoing Ferguson haemorrhoidectomy will be randomly assigned to receive either 2% lidocaine gel or a non-anaesthetic lubricant gel control. Pain scores using a visual analog scale (VAS) will be assessed at 12 and 24 hours, and 2, 3, and 7 days postoperatively. Analgesic consumption will also be measured.

DETAILED DESCRIPTION:
Title: Efficacy of 2% Lidocaine Gel in Reducing Postoperative Pain and Analgesic Consumption Following Haemorrhoidectomy: A Randomized, Double-Blind, Controlled Trial Objective: To assess the effect of 2% lidocaine gel on postoperative pain intensity and analgesic consumption following haemorrhoidectomy.

Study Design: This study is a single-center, randomized, double-blind, controlled trial. Patients will be randomly assigned in a 1:1 ratio to receive either 2% lidocaine gel or a non-anaesthetic water-based lubricant gel (control) using a computer-generated randomization list. The randomization will be stratified by hemorrhoid grade (III or IV). The study medication will be prepared by the hospital pharmacy and provided in identical, pre-filled syringes to ensure blinding of participants and investigators.

Intervention: The intervention group will receive 5 mL of 2% lidocaine gel, while the control group will receive 5 mL of a non-anaesthetic water-based lubricant gel. The study medication will be applied to the perianal region three times per day for 7 days following surgery. Patients will be instructed on the proper application technique and will be provided with a diary to record the time and date of each application.

Outcome Assessment: Postoperative pain will be assessed using a 100 mm visual analog scale (VAS), with 0 representing no pain and 100 representing the worst imaginable pain. Pain scores will be recorded at 12 and 24 hours, and 2, 3, and 7 days after surgery. Patients will also record their analgesic consumption in a diary, including the type, dose, and frequency of analgesics used. Postoperative complications, such as bleeding, infection, or urinary retention, will be assessed by the treating surgeon at each follow-up visit.

Sample Size: A sample size of 222 patients (111 per group) was calculated based on a power of 80%, a significance level of 0.05, and an expected difference in mean VAS scores of 15 mm between the groups, with a standard deviation of 30 mm.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosed with Grade III or IV hemorrhoids
* Candidate for Ferguson haemorrhoidectomy

Exclusion Criteria:

* Not a candidate for Ferguson haemorrhoidectomy
* Recurrent hemorrhoidal disease
* Concurrent anal pathology diagnosed preoperatively, including:
* Anal fistula
* Anal fissure
* Anal polyp
* History of diabetes mellitus
* History of liver cirrhosis
* History of inflammatory bowel disease
* Documented neuropathy
* Coagulation disorders
* Currently on anticoagulants
* Documented allergy to any of the drugs included in the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | Assessed at 12 hours, 24 hours, 2 days, 3 days, and 7 days after surgery
  Postoperative pain measured by Visual Analog Scale (VAS) The Visual Analog Scale (VAS) is a unidimensional measure of pain intensity. Patients mark their pain level on a 10-cm line, where 0 represents "no pain" and 10 represents "the worst pain imaginable". Higher scores indicate greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Chih-I, Study Director — E-DA Hospital
Locations (1):
- E-Da hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The study is a randomized, double-blind, controlled trial evaluating the efficacy of 2% lidocaine gel in reducing postoperative pain and analgesic consumption after haemorrhoidectomy. 222 patients undergoing Ferguson haemorrhoidectomy were randomly assigned to receive either 2% lidocaine gel or a non-anaesthetic lubricant gel control. Pain scores using a visual analog scale (VAS) were assessed at 12 and 24 hours, and 2, 3, and 7 days postoperatively. Analgesic consumption was also measured.
Supporting Information: Study Protocol
Time Frame: 1 year